CLINICAL TRIAL: NCT03072771
Title: A Pilot Trial of Blinatumomab Consolidation Post Autologous Stem Cell Transplantation in Patients With DLBCL
Brief Title: Blinatumomab Consolidation Post Autologous Stem Cell Transplantation in Patients With Diffuse Large B-Cell Lymphoma (DLBCL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201704108
Record Dates: First submitted 2017-03-02; First posted 2017-03-07 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — blinatumomab; Carmustine; Etoposide; Cytarabine; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ASCT + BEAM + Blinatumomab (Experimental): * Standard of care ASCT with BEAM conditioning (carmustine/etoposide/cytarabine/melphalan) - guidelines below, other conditionings are allowed:
    * carmustine is typically given intravenously (IV) at a dose of 300 mg/m^2 on Day -7
    * etoposide is typically given IV at a dose of 100 mg/m^2 twice per day (BID) on Days -6, -5, -4, and -3 (8 doses)
    * cytarabine is typically given IV at a dose of 100 mg/m^2 BID on Days -6, -5, -4, and -3 (8 doses)
    * melphalan is typically given IV at a dose of 140 mg/m*2 on Day -2
  * Auto-SCT will take place on Day 0 as per institutional guidelines
  * Consolidation with blinatumomab will start 6 weeks following auto-SCT. Patients with CR or PR based on pre-transplant PET/CT will receive blinatumomab as a continuous IV infusion (CIVI) at 9μg/day for 1 week, then 28μg/day for 3 weeks (total of 4 weeks).
  Interventions: Drug: Blinatumomab; Procedure: Autologous stem cell transplant; Drug: Carmustine; Drug: Etoposide; Drug: Cytarabine; Drug: Melphalan; Procedure: Peripheral blood draws

INTERVENTIONS:
Drug: Blinatumomab — -Blinatumomab is a bispecific T cell engaging antibody
  Other Names: Blincyto
Procedure: Autologous stem cell transplant — -Standard of care
  Other Names: ASCT; auto-SCT
Drug: Carmustine — -Carmustine is an alkylating agent. It will be sourced from commercial supply. Institutional guidelines will be followed for storage, preparation, and administration of carmustine.
  Other Names: BCNU; BiCNU®
Drug: Etoposide — -Etoposide is a semi-synthetic podophyllotoxin derivative. It will be sourced from commercial supply. Institutional guidelines will be followed for storage, preparation, and administration of etoposide.
  Other Names: VP16
Drug: Cytarabine — -Cytarabine, commonly known as Ara-C, is a synthetic nucleoside. It will be sourced from commercial supply. Institutional guidelines will be followed for storage, preparation, and administration of cytarabine.
  Other Names: Ara-C; Cytosar-U ®; 1-β-Arabinofuranosylcytosine; Arabinosylcytosine; Cytosine arabinoside
Drug: Melphalan — -Melphalan is an alkylating agent. It will be sourced from commercial supply. Institutional guidelines will be followed for storage, preparation, and administration of melphalan.
  Other Names: Alkeran® Tablets; Phenylalanine mustard
Procedure: Peripheral blood draws — -Day +42, Day + 43, Day +56, and Day +100

SUMMARY:
Based on the further need to improve progression-free survival (PFS) and overall survival (OS) post autologous stem cell transplant (SCT) for DLBCL, the hematopoietic profile of patients following auto-SCT, the activity of blinatumomab in DLBCL and its favorable toxicity profile, the investigators propose a pilot study to test blinatumomab as consolidation therapy post auto-SCT for patients with DLBCL.

The investigators hypothesize the blinatumomab consolidation will optimize the effector to target (E-T) ratio and aid in the eradication of remaining tumor cells, leading to decreased relapse and increased overall survival. In addition, since tumor burden will be at a minimum, infusional toxicities including neurologic toxicities may also be limited. The purpose of this pilot study is to study the feasibility and tolerability of blinatumomab consolidation post auto-SCT for patients with chemo-sensitive DLBCL undergoing auto-SCT.

ELIGIBILITY:
Pre-ASCT Inclusion Criteria

* At least 18 years of age
* Histologically confirmed diagnosis of CD19 positive diffuse large B-cell lymphoma (DLBCL) or transformed large cell lymphoma from low grade lymphoma.
* Chemo-sensitive (defined by complete remission (CR) or partial remission (PR) to most recent chemo regimen) based on pre-transplant positron emission tomography (PET) within 2 months of autologous transplant
* Patients with bulky disease are eligible for study provided that the patient not undergo radiation therapy until 30 days after the end of blinatumomab administration.
* Available representative tissue (from fresh or formalin fixed paraffin embedded tissue) from the most recent biopsy or archival tumor tissue for Clonotype evaluation for minimal residual disease (MRD) testing.

Pre-ASCT Exclusion Criteria

* Chemo-resistant (defined by stable disease (SD) or progressive disease (PD) to most recent chemo regimen)
* Pregnant or breastfeeding
* Active central nervous system (CNS) involvement of Non-Hodgkin's Lymphoma (NHL)
* Clinically relevant CNS pathology such as epilepsy, childhood or adult seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis
* Prior stem cell transplant
* Concurrent hematologic or non-hematologic malignancy requiring treatment
* HIV seropositive, or active Hepatitis A, B, or C infection.
* Uncontrolled congestive heart failure (CHF) or other comorbid systemic illnesses or severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.

Eligibility Criteria to Begin Consolidation Therapy

* A participant must meet all of the following criteria on Day +42 visit in order to continue on the study to begin consolidation therapy with blinatumomab.
* Performance status of Eastern Cooperative Oncology Group (ECOG) ≤ 2 or Karnofsky ≥ 60 %
* Absence of clinically relevant CNS pathology such as epilepsy, paresis, aphasia, stroke, sever brain injuries, dementia, or psychosis
* Required clinical laboratory values:

  * Absolute neutrophil count (ANC) ≥ 1,000
  * Platelets ≥ 75,000
  * Hemoglobin ≥ 8 g/dL
  * Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (unless related to Gilbert's or Meulengracht's syndrome)
  * Alkaline phosphatase ≤ 5 x ULN
  * ALT and AST ≤ 5 x ULN
  * Calculated or measured creatinine clearance ≥ 50ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2021-04-07 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Feasibility and tolerability of blinatumomab consolidation post auto-SCT as measured by percentage of patients who can finish a full course of blinatumomab post-auto-SCT | Up to Day 70
  -The primary endpoint is calculated by the proportion of patients who complete a full course of blinatumomab to the total number of patients started blinatumomab after auto-SCT.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 1 year post-auto-SCT
  -PFS is defined as from the date of Day 0 to date of progression or death, which occurs first. They are censored at the last follow-up otherwise.
Progression-free survival (PFS) | 3 years post-auto-SCT
  -PFS is defined as from the date of Day 0 to date of progression or death, which occurs first. They are censored at the last follow-up otherwise.
Overall survival | 1 year post-auto-SCT
  -OS is defined as from the date of Day 0 to date of death. They are censored at the last follow-up otherwise.
Overall survival | 3 years post-auto-SCT
  -OS is defined as from the date of Day 0 to date of death. They are censored at the last follow-up otherwise.
Complete remission rate in patients with residual disease after auto-SCT | Up to Day 100
  -Complete remission=disappearance of all evidence of disease

CONTACTS AND LOCATIONS:
Overall Officials: Armin Ghobadi, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ghobadi A, Foley NC, Cohen J, Rettig MP, Cashen AF, Gehrs L, Christ S, Street E, Wallace N, Ritchey J, Mehta-Shah N, Westervelt P, Fehniger TA, Kahl B, Bartlett NL, DiPersio JF. Blinatumomab consolidation post-autologous stem cell transplantation in patients with diffuse large B-cell lymphoma. Blood Adv. 2024 Feb 13;8(3):513-522. doi: 10.1182/bloodadvances.2023011130. PMID 37871306
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu